CLINICAL TRIAL: NCT03828357
Title: The Evaluation of ICD Defibrillation Systems in a 1.5T Magnetic Resonance Imaging Environment in China
Brief Title: China (CN)_Magnetic Resonance Imaging (MRI)_Implantable Cardiac Defibrillator (ICD) [CN_MRI_ICD]
Acronym: CN_MRI_ICD
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD_930
Record Dates: First submitted 2019-01-08; First posted 2019-02-04 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-03

CONDITIONS: Tachycardia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Ellipse VR with Durata: Ellipse VR single-chamber ICD with a Durata defibrillation lead
  Interventions: Other: Study MRI scan
- Ellipse DR with Durata & Tendril STS: Ellipse DR dual-chamber ICD with a Durata lead in the right ventricle (RV) and a Tendril STS lead in the right atrium (RA).
  Interventions: Other: Study MRI scan
- Ellipse DR with Optisure and Isoflex: Ellipse DR dual-chamber ICD with an Optisure defibrillation lead in the right ventricle (RV) and an Isoflex lead in the right atrium (RA).
  Interventions: Other: Study MRI scan
- Quadra Assura MP CRT-D: Quadra Assura MP CRT-D with an Optisure or Durata defibrillation lead in the RV, an Isoflex or Tendril STS lead in the RA, and a Quartet lead in the LV
  Interventions: Other: Study MRI scan

INTERVENTIONS:
Other: Study MRI scan — At least forty-five (45) days after system implantation or after a system revision, Subjects will undergo a study-related MRI scan at 1.5T.

SUMMARY:
This clinical study is to evaluate the safety and effectiveness of the Ellipse VR/DR implantable cardiac defibrillators (ICDs) and the Quadra Assura MP cardiac resynchronization therapy defibrillators (CRT-Ds), with Durata or Optisure defibrillation leads, Tendril STS or Isoflex pacing leads, and the Quartet quadripolar leads in a 1.5T MRI environment for MR-conditional labeling expansion of these market-approved ICD/CRT-D systems in China.

Note: Protocol updated: Fortify Assura VR/DR ICD removed; Quadra Assura MP CRT-D and Quartet leads added. The Detailed Description Section below was updated upon protocol amendment.

DETAILED DESCRIPTION:
Endpoints, and contents of clinical study

Objectives:

The objective of this clinical study is to evaluate the safety and effectiveness of the Ellipse VR/DR implantable cardiac defibrillators (ICDs) and the Quadra Assura MP cardiac resynchronization therapy defibrillators (CRT-Ds), with Durata or Optisure defibrillation leads, Tendril STS or Isoflex pacing leads, and the Quartet quadripolar leads in a 1.5T MRI environment for MR-conditional labeling expansion of these market-approved ICD/CRT-D systems in China.

There are four device combination groups in this clinical study as outlined below:

* Group 1: Ellipse VR single-chamber ICD with a Durata lead in the right ventricle (RV).
* Group 2: Ellipse DR dual-chamber ICD, with a Durata lead in the RV and a Tendril STS lead in the right atrium (RA).
* Group 3: Ellipse DR dual-chamber ICD with a Optisure lead in the RV and a Isoflex lead in the RA.
* Group 4: Quadra Assura MP CRT-D with a Durata or Optisure lead in the RV, a Tendril STS or Isoflex lead in the RA, and a Quartet lead in the left ventricle (LV).

Endpoints

Primary Endpoints

* Safety: Freedom from MRI-scan related complications related to the ICD device and/or leads from the time of the MRI scan to 1-month post-MRI scan testing.
* Effectiveness: Proportion of leads with a capture threshold increase of ≤ 0.5V at 0.5ms for RA and RV leads and ≤1.0V at 0.5ms for LV leads from pre-MRI scan to 1-month post-MRI scan testing.
* Effectiveness: Proportion of leads with a sensing amplitude decrease of ≤ 50% from pre-MRI scan testing to 1-month post-MRI scan.

Descriptive Endpoint(s)

Descriptive endpoints are reported using only summary statistics and no hypothesis tests will be performed.

The following data will be collected:

1. Demographics: gender, age, ethnicity, race, cardiac disease history, arrhythmia history, indication for ICD implant, history of smoking, etc.
2. Device electrical measurements at the MRI Scan Visit (pre- and post-scan) and at the 1 Month Post Scan Visit
3. ADE, SADE, USADE
4. Mortality
5. Number of non-study MRI scans
6. Summarize number of subjects that returned to usual programming after the MRI scan and number of subjects, if any, experiencing delays in reprogramming

This is a prospective, multi-center, single-arm study to evaluate the safety and effectiveness of the Ellipse VR/DR ICDs, and the Quadra Assura MP CRT-D, with Durata or Optisure defibrillation leads, Tendril STS or Isoflex pacing leads, and the Quartet quadripolar LV lead in a 1.5T MRI environment for MR-conditional labeling expansion in China.

This study will be conducted in at least 6 centers in China and at least 60 subjects who provide consent for participation will be enrolled. Subjects will be considered enrolled after providing consent. Subjects will be implanted with any one of the device/lead combination groups outlined in Figure 1, depending on their clinical need as determined by the Investigators. At least 15 subjects will be enrolled in each group.

* Group 1 will have at least 15 enrolled subjects with the Ellipse VR single-chamber ICD with a Durata lead in the RV.
* Group 2 will have at least 15 enrolled subjects with the Ellipse DR dual-chamber ICD with a Durata lead in the RV and a Tendril STS lead in the RA.
* Group 3 will have at least 15 enrolled subjects with the Ellipse DR dual-chamber ICD with a Optisure lead in the RV and a Isoflex lead in the RA.
* Group 4 will have at least 15 enrolled subjects with a Quadra Assura MP CRT-D and an Optisure or Durata lead in the RV, an Isoflex or Tendril STS lead in the RA, and a Quartet lead in the LV.

The enrollment group and group 4 lead pairing will be at the discretion of the Investigator, dependent on patient needs in conjunction with study needs to fulfill study goals.

At least forty-five (45) days after system implantation or after a system revision, subjects will have a baseline visit followed by an MRI visit; subjects will undergo a study-related MRI scan at 1.5T. Subjects will have a 1-month follow-up after the study MRI scan. The minimum duration of each subject's participation is approximately 2.5 months from enrollment. The expected duration of enrollment is approximately 14 months. The total duration of clinical study is expected to be 16.5 months.

The study population includes male and female Chinese nationals that meet the eligibility requirements and give consent for the study. Vulnerable subjects, such as minors or those unable to provide consent are excluded from participating.

Inclusion criteria

Assessment for general eligibility criteria is based on medical records of the site and interview with a candidate patient. If some of the clinical and laboratory tests are not included in site standard tests, they must be done but after written informed consent is obtained. Patients must meet ALL the inclusion criteria to be considered for the clinical study. If ANY of the exclusion criteria are met, the patient is excluded from the clinical study and cannot be enrolled.

To participate in this clinical study, the subject must meet all the following inclusion criteria:

* Have an approved indication for implantation of an ICD, or CRT-D
* Be a Chinese national
* Will be implanted with one of the following device/lead combinations evaluated in this study:

  * Group 1: Ellipse VR single-chamber ICD with a Durata lead in the RV
  * Group 2: Ellipse DR dual-chamber ICD, with a Durata lead in the RV and a Tendril STS lead in the RA
  * Group 3: Ellipse DR dual-chamber ICD with a Optisure lead in the RV and a Isoflex lead in the RA
  * Group 4: Quadra Assura MP CRT-D and an Optisure or Durata lead in the RV, an Isoflex or Tendril STS lead in the RA, and a Quartet lead in the LV
* Be willing to undergo an elective MRI scan without sedation ≥ 45 days after implant NOTE: Antianxiety agents (e.g. minor tranquilizers, etc.) may be used as long as the patient can communicate with site personnel during the MRI scan
* Be able to provide informed consent for study participation (legal guardian or legally authorized representative is NOT acceptable)
* Be willing and able to comply with the prescribed follow-up tests and procedures
* Are not contraindicated for an MRI scan (per the MRI Screening Form)
* Subjects who are at least 18 years of age (or older, required by local law)

Exclusion criteria

Subjects who meet any of the following exclusion criteria must be excluded from the clinical investigation:

* Have a competitor's MRI compatible endocardial lead implanted or capped
* Have another existing active implanted medical device, e.g., neurostimulator, infusion pump, etc. that has MR labeling that will not allow the MRI scans per this protocol to be completed.
* Have other non-MRI compatible device or material implanted. The following examples may be included as long as labelling of these devices allow MRI scans conducted per this protocol:

  * MRI compatible knee replacements, hip replacements, stents, etc.
  * MRI compatible mechanical, prosthetic, and bio prosthetic heart valves
  * Non-removable dental implants
* Have a lead extender, adaptor, or capped/abandoned lead
* Enrolled or intend to participate in a clinical drug and/or device study (investigational device, investigational drug, new indication for a device or drug or additional testing beyond standard of care procedures), which could confound the results of this study as determined by Abbott.
* Pregnant or planning to become pregnant during the duration of the subject's participation in the study
* Have a life expectancy of less than 12 months due to any condition

Effectiveness evaluation method

There are two effectiveness endpoints to be evaluated in this study.

1. Description of the effectiveness endpoints

   * Proportion of leads with a capture threshold increase of ≤ 0.5V at 0.5ms for RA and RV leads and ≤ 1.0V at 0.5ms for LV leads from pre-MRI scan to 1-month post-MRI scan testing.
   * Proportion leads with a sensing amplitude decrease of ≤ 50% from pre-MRI scan testing to 1-month post-MRI scan.
2. Selection of method and time for evaluation, recording and analysis of the effectiveness endpoints Since the objective is to evaluate the effect of MRI exposure for the ICD/ CRT-D device groups included in this study, the effectiveness parameters were selected to compare abnormal changes in device performance from pre- to 1-month post- MRI scan. The pre-MRI measurements are collected within the same day prior to the MRI scan. The 1-month post-MRI scan measurements are collected at 30 days post-MRI scan (within +14 days) to ensure any effect of the MRI exposure is captured.

The effectiveness parameters are recorded directly from the device. The device measurements will be obtained using the Merlin programmer to interrogate the device during study visits. The analysis of the effectiveness parameters will be conducted on all subjects with complete data from pre- to 1-month post-MRI scan.

Safety evaluation method There is one safety primary endpoint to be evaluated in this study.

1. Description of the safety endpoint Freedom from MRI-scan related complications from the time of the MRI scan to 1-month post-MRI scan testing.
2. Selection of method and time for evaluation, recording and analysis of the safety endpoints Since the objective is to evaluate the effect of MRI exposure for the ICD/ CRT-D device groups included in this study, the safety parameters were selected to include only MRI-scan related complications from the time of device programming for an MRI scan to 1-month post-MRI scan. An independent physician CEC will adjudicate all adverse device effects during this period to determine the relatedness to the MRI scan.

Safety surveillance within this study and the safety reporting, both performed by the investigator, starts as soon as the subject completes the pre-MRI visit testing and the MRI Settings have been programmed according to the protocol. The safety surveillance and the safety reporting will continue until the last study visit has been performed, the subject is deceased, the subject/investigator concludes his participation into the clinical study or the subject withdrawal from the clinical study.

Monitoring plan

Sponsor and/or designee will monitor the clinical study over its duration according to the CIP-specific monitoring plan which will include the planned extent of source data verification.

Prior to initiating any procedure, the Sponsor monitor (or delegate) will ensure that the following criteria are met:

* The investigator understands and accepts the obligation to conduct the clinical study according to the CIP and applicable regulations, and has signed the Clinical Trial Agreement.
* The Investigator and his/her staff should have sufficient time and facilities to conduct the clinical study and should have access to an adequate number of appropriate subjects to conduct the clinical study.
* Source documentation (including original medical records) must be available to substantiate proper informed consent procedures, adherence to CIP procedures, adequate reporting and follow-up of adverse events, accuracy of data collected on case report forms, and device information.
* The Investigator/site will permit access to such records. A monitoring visit sign-in log will be maintained at the site. The Investigator will agree to dedicate an adequate amount of time to the monitoring process. The Investigator and/or research coordinator will be available for monitoring visits. It is expected that the Investigator will provide the monitor with a suitable working environment for review of clinical study-related documents.

Statistical considerations

This study is an observational study to meet the requirements for device approval by the National Medical Products Administration (NMPA, previously China FDA). There is no endpoint hypotheses testing planned in this study. The endpoints, demographics, safety and device data will be summarized using descriptive statistics as outlined in the Statistical Analysis Plan (SAP).

Any major changes to the SAP will be documented in an amendment to the SAP. Less significant changes to the planned analyses will be documented in the final report(s).

Data management

Study data will be handled according to China Device GCP (Order 25). The Leading PI and his/her associated organization (leading Unit) will be responsible for compiling and submitting all required reports to governmental agencies.

Before the submission, Leading PI and his/her associated organization (leading Unit) should allow sponsor to have a copy of the above reports for reviewing, and providing comments for Leading PI and his/her associated organization consideration.

Data will be analyzed by the Leading PI and his/her associated organization (leading Unit) and/or its affiliates. The Leading PI and his/her associated organization (leading Unit)'s also agree that data may be transferred to the Sponsor's locations worldwide and/or any other worldwide regulatory authority in support of a market-approval application.

ELIGIBILITY:
Inclusion Criteria:

To participate in this clinical study, the subject must meet all of the following inclusion criteria:

* Have an approved indication for implantation of a ICD
* Be a Chinese national
* Will be implanted with one of the following device/lead combinations evaluated in this study:

  * Group 1: Ellipse VR single-chamber ICD with a Durata lead in the right ventricle (RV)
  * Group 2: Fortify Assura single-chamber ICD, with an Optisure lead
  * Group 3: Ellipse DR dual-chamber ICD with a Durata lead in the RV and a Tendril STS lead in the right atrium (RA)
  * Group 4: Fortify Assura ICD and an Optisure lead in the RV and an Isoflex lead in the RA
* Be willing to undergo an elective MRI scan without sedation ≥ 45 days after implant NOTE: Antianxiety agents (e.g. minor tranquilizers, etc.) may be used as long as the patient can communicate with site personnel during the MRI scan
* Be able to provide informed consent for study participation (legal guardian or legally authorized representative is NOT acceptable)
* Be willing and able to comply with the prescribed follow-up tests and procedures
* Are not contraindicated for an MRI scan (per the MRI Screening Form)
* Subjects who are at least 18 years of age (or older, required by local law)

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria must be excluded from the clinical investigation:

* Have a competitor's MRI compatible endocardial lead implanted or capped
* Have another existing active implanted medical device, e.g., neurostimulator, infusion pump, etc. that has MR labeling that will not allow the MRI scans per this protocol to be completed.
* Have other non-MRI compatible device or material implanted. The following examples may be included as long as labelling of these devices allow MRI scans conducted per this protocol:

  * MRI compatible knee replacements, hip replacements, stents, etc.
  * MRI compatible mechanical, prosthetic, and bio prosthetic heart valves
  * Non-removable dental implants
* Have a lead extender, adaptor, or capped/abandoned lead
* Enrolled or intend to participate in a clinical drug and/or device study (investigational device, investigational drug, new indication for a device or drug or additional testing beyond standard of care procedures), which could confound the results of this study as determined by Abbott.
* Pregnant or planning to become pregnant during the duration of the subject's participation in the study
* Have a life expectancy of less than 12 months due to any condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes male and female Chinese nationals that meet the eligibility requirements and give consent for the study. Vulnerable subjects, such as minors or those unable to provide consent are excluded from participating.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ellipse VR With Durata | Ellipse DR With Durata & Tendril STS | Ellipse DR With Optisure and Isoflex | Quadra Assura MP CRT-D
Started | 15 | 15 | 15 | 15
Completed | 14 | 14 | 15 | 12
Not Completed | 1 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Population: All consented subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Ellipse VR With Durata | Ellipse DR With Durata & Tendril STS | Ellipse DR With Optisure and Isoflex | Quadra Assura MP CRT-D | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (9.9) | 61.5 (13.4) | 58.9 (14) | 57.7 (10.1) | 58.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 8 | 10 | 39
  Male | 2 | 7 | 7 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 15 | 14 | 15 | 15 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 15 | 15 | 15 | 15 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 15 | 15 | 15 | 15 | 15
Cardiovascular History- dominant type of cardiomyopathy [Count of Participants; unit: Participants]
  Non-ischemic | 10 | 6 | 7 | 11 | 34
  Ischemic | 1 | 4 | 6 | 1 | 12
  None | 4 | 5 | 2 | 3 | 14
Prior Cardiac Interventions [Count of Participants; unit: Participants]
  PTCA/ Stents/ Atherectomy | 1 | 3 | 5 | 1 | 10
  Ablation | 1 | 2 | 1 | 0 | 4
  none | 13 | 10 | 9 | 14 | 46
Arrhythmia History [Count of Participants; unit: Participants]
  Ventricular | 4 | 7 | 10 | 2 | 23
  Non-ventricular | 5 | 1 | 3 | 2 | 11
  Other or not recorded | 6 | 7 | 2 | 11 | 26
Primary Indication for ICD/CRT Implant [Count of Participants; unit: Participants]
  Cardiac Arrest | 1 | 0 | 0 | 0 | 1
  Ventricular Tachycardia | 2 | 7 | 5 | 0 | 14
  Ischemic Cardiomyopathy | 1 | 4 | 4 | 0 | 9
  Non-ischemic Cardiomyopathy | 10 | 3 | 3 | 0 | 16
  Familial Condition | 1 | 1 | 0 | 0 | 2
  Syncope | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 2 | 0 | 2
  HF with wide QRS | 0 | 0 | 0 | 14 | 14
  Reduced EF with frequent dependence on V-pacing | 0 | 0 | 0 | 1 | 1
History of Smoking [Count of Participants; unit: Participants]
  Yes | 10 | 7 | 6 | 4 | 27
  No | 5 | 8 | 9 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From Magnetic Resonance Imaging (MRI) Scan Related Complications
Description: Freedom from Magnetic Resonance Imaging (MRI) scan related complications related to the Implantable Cardiac Difibrillator (ICD) device and/or leads from the time of the MRI scan to 1-month post-MRI scan testing.
Time Frame: 1 month from MRI scan
Population: The primary safety endpoint analysis is conducted on subjects in the Analysis Cohort who completed the 1-month post-MRI scan visit or have MRI-scan related complication(s) related to the ICD/CRT-D device and/or leads.
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipse VR With Durata | Ellipse DR With Durata & Tendril STS | Ellipse DR With Optisure and Isoflex | Quadra Assura MP CRT-D
Number analyzed (Participants) | 14 | 14 | 15 | 12
Participants | 14 | 14 | 15 | 12

2. Primary Outcome: Effectiveness Outcomes: Percentage of Leads With a Capture Threshold Increase
Description: Proportion of leads with a capture threshold increase of ≤ 0.5V at 0.5ms from pre-MRI scan to 1-month post-MRI scan testing.
Time Frame: pre-MRI scan to 1 month post-MRI scan
Population: The primary analysis for the primary effectiveness endpoint #1 is conducted on subjects in the Analysis Cohort who have completed the 1-month post-MRI scan visit, with evaluable device data available for analysis and meet all the following criteria:
  1. Have pre-MRI scan visit data for capture threshold
  2. Have 1-month post-MRI scan visit data for capture threshold
  3. Have not undergone any lead repositioning or replacement since the MRI scan up to 1-month post-MRI scan.
Measure: Number; unit: percentage of leads meeting criteria
Units Other Than Participants: leads
Arm/Group | Ellipse VR With Durata | Ellipse DR With Durata & Tendril STS | Ellipse DR With Optisure and Isoflex | Quadra Assura MP CRT-D
Number analyzed (Participants) | 14 | 14 | 14 | 12
Number analyzed (leads) | 14 | 28 | 28 | 36
percentage of leads meeting criteria
  Right Atrial (RA) leads | NA — no RA leads in this group | 100 | 100 | 100
  Right Ventricular (RV) leads | 100 | 100 | 100 | 100
  Left Ventricular (LV) leads | NA — no LV leads in this group | NA — no LV leads in this group | NA — no LV leads in this group | 100

3. Primary Outcome: The Percentage of Leads With a Sensing Amplitude Decrease of ≤ 50% From Pre-MRI Scan Testing to 1-month Post-MRI Scan.
Description: Proportion of subjects with a sensing amplitude decrease ≤ 50% from pre-MRI scan to 1-month post MRI scan % (n/N)
Time Frame: pre-MRI scan to 1 month post-MRI scan
Population: The primary analysis for the primary effectiveness endpoint #2 is conducted on subjects in the Analysis Cohort who undergo the 1-month post-MRI scan testing, with evaluable device data available for analysis to be performed, and meet all the following criteria:
  1. Have pre-MRI scan visit data for sensing amplitude
  2. Have 1-month post-MRI scan visit data for sensing amplitude
  3. Have not undergone any ICD/CRT-D lead repositioning or replacement since the MRI scan up to 1-month post-MRI scan.
Measure: Number; unit: percentage of leads meeting criteria
Units Other Than Participants: leads
Arm/Group | Ellipse VR With Durata | Ellipse DR With Durata & Tendril STS | Ellipse DR With Optisure and Isoflex | Quadra Assura MP CRT-D
Number analyzed (Participants) | 14 | 14 | 14 | 12
Number analyzed (leads) | 14 | 28 | 28 | 36
percentage of leads meeting criteria
  Right Atrial Leads | NA — no Right Atrial Leads in this group | 100 | 100 | 92
  Right Ventricular Leads | 100 | 100 | 100 | 100

4. Secondary Outcome: Device Electrical Measurements
Description: Summaries of electrical measurements taken in the Analysis Cohort at Pre-MRI scan, Post-MRI scan, and 1-month post MRI scan. The stable electrical measurements from pre-MRI scan to post-MRI scan and 1-month post MRI scan indicate that the MRI scan did not impact the electrical performance of the Ellipse ICD or Quadra Assura CRT-D system
Time Frame: Pre-MRI scan, Post MRI scan, 1 month follow-up
Population: patients that had respective electrical measurements captured at pre-MRI, post-MRI or 1-month follow-up
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Ellipse VR With Durata | Ellipse DR With Durata & Tendril STS | Ellipse DR With Optisure and Isoflex | Quadra Assura MP CRT-D
Number analyzed (Participants) | 15 | 14 | 15 | 14
Volts
  pre-MRI: Right ventricular capture threshold | 0.72 (0.19) | 0.75 (0.24) | 0.80 (0.19) | 0.7 (0.22)
  pre-MRI: Right ventricular sensing amplitude | 0.0113 (0.0015) | 0.0110 (0.0021) | 0.0108 (0.0019) | 0.0119 (0.2)
  post-MRI: Right ventricular capture threshold | 0.71 (0.19) | 0.75 (0.20) | 0.73 (0.18) | 0.63 (0.17)
  post-MRI: Right ventricular sensing amplitude | 0.0112 (0.0017) | 0.0113 (0.0022) | 0.0108 (0.0017) | 0.0117 (0.0008)
  1 month follow-up: Right ventricular capture threshold | 0.73 (0.18) | 0.73 (0.18) | 0.80 (0.2) | 0.63 (0.2)
  1 month follow-up: Right ventricular sensing amplitude | 0.0114 (0.0014) | 0.0109 (0.0026) | 0.0112 (0.0013) | 0.0117 (0.0007)

5. Secondary Outcome: Number of Participants With Whole Body (WB) SAR Values Measured ≥ 1.8 W/kg
Description: Whole body (WB) SAR values from the RF intensive MRI scans.
  Abbott is seeking MR-conditional labeling for MRI scans in Normal Operating Mode (WB Specific Absorption Rate (SAR) up to 2 W/kg). Achieving a WB SAR of exactly 2 W/kg is not feasible since the MR technologist must adjust multiple interdependent scab parameters to increase the WB SAR. Therefore, an acceptable limit of ≥ 1.8 W/kg (within 10%) was established as part of the MRI scan sequence guideline document for this study prior to site enrollments to account for expected user variability.
Time Frame: during MRI scan
Population: Subjects that completed study MRI scan were included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipse VR With Durata | Ellipse DR With Durata & Tendril STS | Ellipse DR With Optisure and Isoflex | Quadra Assura MP CRT-D
Number analyzed (Participants) | 14 | 14 | 15 | 12
Participants | 14 | 13 | 13 | 12

6. Secondary Outcome: Summary of Subjects That Returned to Usual Programming
Description: Subjects that returned to usual programming after the MRI scan and the number of subjects experiencing delays in disabling MRI settings after the MRI scan
Time Frame: MRI scan visit
Population: Subjects that completed MRI scan were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipse VR With Durata | Ellipse DR With Durata & Tendril STS | Ellipse DR With Optisure and Isoflex | Quadra Assura MP CRT-D
Number analyzed (Participants) | 14 | 14 | 15 | 12
Participants
  Number of subjects that returned to usual programming after the MRI scan | 14 | 14 | 15 | 12
  Number of subjects with a delay in disabling MRI settings after MRI scan | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: from the period between device programming of MRI settings to 1-month post-MRI scan, as defined in the protocol.
Arm/Group | Ellipse VR With Durata | Ellipse DR With Durata & Tendril STS | Ellipse DR With Optisure and Isoflex | Quadra Assura MP CRT-D
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/15 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/14 | 3/14 | 2/15 | 1/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 1/15 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ellipse VR With Durata (N=14) | Ellipse DR With Durata & Tendril STS (N=14) | Ellipse DR With Optisure and Isoflex (N=15) | Quadra Assura MP CRT-D (N=12)
OTHER: CERVICAL SPONDYLOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER:HEART FAILURE (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER:Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER: CAROTID SCLEROSIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER: HYPERKALEMIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER: DILATED CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER:INAPPROPIATE SHOCK (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ellipse VR With Durata (N=14) | Ellipse DR With Durata & Tendril STS (N=14) | Ellipse DR With Optisure and Isoflex (N=15) | Quadra Assura MP CRT-D (N=12)
OTHER: VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT03828357/Prot_SAP_000.pdf